CLINICAL TRIAL: NCT06337305
Title: Resiliency in Patients Undergoing Radical Cystectomy for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Lee, MD, Associate Professor and Urologic Oncology Fellowship Director, University of Kansas Medical Center
Other Study IDs: STUDY00146138
Record Dates: First submitted 2024-03-08; First posted 2024-03-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder cancer patients undergoing radical cystectomy.: This is a prospective cross-sectional survey of bladder cancer patients undergoing radical cystectomy.

SUMMARY:
This is a prospective cross-sectional survey-based study composed of both a retrospective chart review and 3-series patient survey. This study will help elicit potential areas throughout the perioperative course of radical cystectomy to improve patient resilience and quality of life, providing opportunity for future interventional studies.

DETAILED DESCRIPTION:
This is a prospective cross-sectional survey-based study composed of both a retrospective chart review and 3-series patient survey. This study will help elicit potential areas throughout the perioperative course of radical cystectomy to improve patient resilience and quality of life, providing opportunity for future interventional studies. Primarily, the study will evaluate health related quality of life and resiliency in patients throughout the perioperative course of a radical cystectomy for bladder cancer.

The primary objective will be the correlation of the Connor-Davidson Resilience Scale (CD-RISC-25) and the Functional Assessment of Cancer Therapy-Bladder-Cystectomy (FACT-BL-Cys) score.

Patients will be identified and undergo consent and baseline assessments, including completion of surveys prior to their cystectomy. A retrospective chart review will also be completed to record information regarding patient's cancer stage, treatment status, diagnosis date, insurance type, and related medical conditions and medications. Data from retrospective chart review will be collected and recorded in a secure REDCap database for all eligible patients.

Subsequent surveys will be administered again at approximately 10-30 days postoperatively, as well as 60-120 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of bladder cancer
* Patients electing to undergo radical cystectomy as treatment
* ≥ 18 years of age
* Able to speak and read English
* Willing and able to provide informed consent
* Functioning telephone number or access to one

Exclusion Criteria:

* Patients opting to not undergo radical cystectomy
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radical cystectomy for bladder cancer
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2023-08-19 (Actual)

PRIMARY OUTCOMES:
Change in resiliency as measured by the Connor-Davidson Resilience Scale (CD-RISC-25). | Prior to radical cystectomy, 10-30-days post-operative, and 90-days (+/-30-days) post-operative
  The Connor-Davidson Resilience scale is a 25-item self-administered instrument for assessing resilience that is consistent in a variety of populations, including clinical and community.
  Scoring: 0-100 (sum total of all items, each of which is scored 0-4). Higher score reflects greater resilience.
Change in quality of life in patients undergoing radical cystectomy as measured by the Functional Assessment of Cancer Therapy-Bladder-Cystectomy (FACT-Bl-Cys). | Prior to radical cystectomy, 10-30-days post-operative, and 90-days (+/-30-days) post-operative
  The FACT-BL-Cys is a condition-specific instrument for patients undergoing radical cystectomy to measure quality of life.
  Scoring: 0-168 (sum total of all items). Higher score reflects better health-related quality of life.
Change in quality of life in patients undergoing radical cystectomy as measured by the PROMIS-29. | Prior to radical cystectomy, 10-30-days post-operative, and 90-days (+/-30-days) post-operative
  The PROMIS-29 is a disease non-specific measure of pain intensity using a 1-5 rating and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance).
  Scoring: High scores mean more of the concept being measured.

SECONDARY OUTCOMES:
Identification of clinical and demographic factors in bladder cancer patients | Baseline to 90-days (+/-30 days) post-operative
  Identify clinical and demographic factors related to higher post-cystectomy resiliency in patients with bladder cancer.
Demographics | Baseline to 90-days (+/-30 days) post-operative
  Characterize trends that correspond with greater levels of resiliency and quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No